CLINICAL TRIAL: NCT05594316
Title: Efficacy of Trichloroacetic Acid in Patients of Alopecia Areata : Clinico-histopathological Study
Brief Title: New Treatment of Alopecia Areata
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hossam Mamdouh Anter Esmail, Assisstant lecturer of dermatology,venerology and andrology, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hossam pulse
Record Dates: First submitted 2022-10-19; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Alopecia Areata
Keywords: alopecia areata AA
MeSH Terms: conditions — Alopecia Areata | interventions — Trichloroacetic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single group (Other): Trichloroacetic acid
  Interventions: Drug: Trichloroacetic acid

INTERVENTIONS:
Drug: Trichloroacetic acid — 5. Patients will be subjected to 3 session of trichloroacetic acid 35% one month apart.

SUMMARY:
Abstract: Alopecia areata is believed to be an autoimmune disease resulting from a breach in the immune privilege of the hair follicles causing non scarring hair loss.

Methods: our study included 40 patients from may 2019 to july 2022 diagnosed clinically, dermatoscopically and pathologically as alopecia areata Data were enrolled from department of dermatology and venereology, Al-Hussein hospital.

DETAILED DESCRIPTION:
For each patient the following will be done :

1. History taking including ( age, sex, disease duration, family history, history of drug intake, smoking and history of any associated disease ).
2. All patients will give a written, informed consent for induction.
3. Basic photographs will be taken to assess site, size (by cm), number, Extent of the patch using D5300 camera with lens (18-55).
4. Patients will be subjected to 3 session of trichloroacetic acid (TCA) 35% one month apart.
5. serial photographs and dermoscopic examination every month will be done and patient will be score.
6. Efficacy will be assessed using prognostic scoring system for density, pigmentation, and texture of growing hair.
7. histopathological examination will be done before the first session and one month after third session.

ELIGIBILITY:
Inclusion Criteria:

* Alopecia areata multilocularis and alopecia totalis. Age from 16-60 years old. Ophiasis pattern alopecia areata.

Exclusion Criteria:

* Age less than 16 and more than 60years old. Alopecia areata of the face.
* Patient under treatment.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Mac Donald Hull and Norris grading system | 4 weeks after the end of treatment
  regrowth of vellus hair, regrowth of sparse pigmented terminal hair, regrowth of terminal hair with patches of alopecia and regrowth of terminal hair on scalp.
Scoring of texture of regrown hair | after each session and 4 weeks after the end of treatment
  Fine vellus hair, Intermediate hair,Normal coarse hair
Scoring of pigmentation of regrown hair | after each session and 4 weeks after the end of treatment
  Partially pigmented, Moderately pigmented, Normally pigmented
Scoring for density of hair regrowth | after each session and 4 weeks after the end of treatment
  No hair growth, 1%-25% growth, 26%-50% growth, 51%-75% growth and 76%-100% growth
Scoring of overall response at the end of the study | after each session and 4 weeks after the end of treatment
  No response, Minimal response, Moderate response, Good response and Excellent response
histopathological changes | after each session and 4 weeks after the end of treatment
  appearance of lymphocytes around hair follicle, appearance of new blood vessels and size of thickness of hair follicles
trichoscopic parameters | after each session and 4 weeks after the end of treatment
  determine exclamation mark hairs, black dots, yellow dots and broken hairs

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Al-Azhar university, faculty of medicine, Cairo
  - Al-Azhar university, Cairo

IPD SHARING:
Plan to Share IPD: Undecided